CLINICAL TRIAL: NCT05047224
Title: Addressing Disparities in ASD Diagnosis Using a Direct-to-home Telemedicine Tool: Evaluation of Diagnostic Accuracy, Psychometric Properties, and Family Engagement
Brief Title: Addressing Disparities in Autism Spectrum Disorder Diagnosis Using a Direct-to-home Telemedicine Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Zachary Warren, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 210760; 1R01MH127228-01 (NIH)
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; tele-assessment
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Clinicians conducting in-person diagnostic evaluations will be blind to the outcomes of initial telehealth diagnostic appointments until after in-person assessments are administered and scored. Clinicians will be unblinded to telehealth diagnostic outcomes prior to sharing the results of in-person assessment with families.
  Clinicians conducting the second telehealth appointments for test-retest and interrater reliability purposes will be blind to recruitment pathway and diagnostic outcome from the initial telehealth appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-assessment + in-person assessment (Experimental): Participants in this group will receive a tele-assessment using the TAP and will attend a traditional, in-person evaluation for autism spectrum disorder in a clinic setting.
  Interventions: Behavioral: Tele-assessment + in-person assessment
- Tele-assessment only (Active Comparator): Participants in this group will receive a tele-assessment using the TAP, followed by a second, shorter tele-assessment.
  Interventions: Behavioral: Tele-assessment only

INTERVENTIONS:
Behavioral: Tele-assessment + in-person assessment — Participants will complete a tele-assessment using the TAP. They will complete a traditional, in-person autism spectrum disorder assessment approximately two weeks later.
  Arms: Tele-assessment + in-person assessment
Behavioral: Tele-assessment only — Participants will complete a tele-assessment using the TAP. They will complete a second, shorter tele-assessment approximately two weeks later.
  Arms: Tele-assessment only

SUMMARY:
The investigators propose to evaluate the use of a telemedicine tool, the TELE-ASD-PEDS (TAP), that is designed to assess for autism spectrum disorder (ASD) symptoms in toddlers. The TAP was developed at VUMC by a team of clinical psychologists with expertise in the early identification of ASD. The TAP has been studied in controlled laboratory settings, with high levels of family and clinician satisfaction, as well as excellent agreement with blinded comprehensive ASD evaluation. The TAP has also been used to complete direct-to-home telemedicine assessments during the COVID-19 pandemic. However, the investigators have not yet compared direct-to-home assessments using the TAP with gold standard, in-person ASD assessments. It has also not yet been studied in a diverse sample of families or with providers outside of VUMC. This study will allow the investigators to address those gaps.

DETAILED DESCRIPTION:
The investigators propose to evaluate the use of a telemedicine tool, the TELE-ASD-PEDS (TAP), that is designed to assess for autism spectrum disorder (ASD) symptoms in toddlers. This study will recruit 360 toddlers (18-42 months of age) across two sites (VUMC and the University of California, Davis). All toddlers will receive in-home telemedicine assessment for ASD using the TAP. This study has two aims. The first aim will randomize participants to receive either (1) telemedicine assessment and an in-person ASD assessment or (2) telemedicine-based assessment only. The investigators will measure diagnostic accuracy of the TAP in comparison to gold standard, in-person ASD assessment. The investigators will also assess test-retest reliability, inter-rater reliability, and the sensitivity, specificity, and positive predictive value of the TAP. In the second aim, all 360 families will be followed over six months to evaluate service access, family engagement, and family perceptions of the diagnostic process.

ELIGIBILITY:
Inclusion Criteria for Children:

* Child between 18 and 42 months of age
* Child and primary caregiver live within a 3-hour driving radius of one of the sites (i.e., VUMC or UC Davis)

Inclusion Criteria for Caregivers:

* Age 18 years or older
* Parent or legal guardian of participating child
* Has access to technology (e.g., phone, laptop, or tablet with internet connection and audio-visual capabilities) to connect to the tele-assessment platform
* Sufficient facility with English to participate in the procedures and complete study measures.

Exclusion Criteria for Children:

* Severe sensorimotor impairment that cannot be corrected and would interfere with completion of study activities
* Medical conditions for which tele-evaluation of ASD symptoms is likely to be inappropriate or complex (i.e., rare genetic syndromes, severe epilepsy, fragile health).

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the TAP | Baseline to completion of in-person autism evaluation, approximately two weeks
  The investigators will compare diagnoses made from the tele-assessment using TAP to those from in-person evaluation. We will calculate the percent agreement between diagnoses assigned in each condition.
Validity of the TAP | Baseline to completion of in-person autism evaluation, approximately two weeks
  Validity of the TAP will be measured by assessing the psychometric properties of the tool. Estimated performance metrics will include positive predictive value (PPV), negative predictive value (NPV), sensitivity, and specificity of the TAP.

SECONDARY OUTCOMES:
Family perceptions of tele-assessment | Baseline
  Family perceptions of tele-assessment will be measured by the Parent Perceptions of Telemedicine (PPT) survey. The PPT is an 11-question survey. Seven questions are measured on a three-point scale and will provide quantitative data. Each question ranges from 1 (not true) to 3 (very true). Possible survey scores can range from 7 to 21. Higher scores indicate more positive perceptions of tele-assessment.
Family satisfaction with diagnostic services | Baseline and six-month follow-up
  Family satisfaction with diagnostic services will be measured by the Parent Service Satisfaction (PSS) survey. The PSS is an 7-question survey. Questions are measured on a three-point scale ranging from 1 (not true) to 3 (very true). Possible survey scores can range from 7 to 21. Higher scores indicate higher satisfaction with diagnostic services.
Family empowerment | Baseline and six-month follow-up
  Family empowerment will be measured using the Family Empowerment Scale (FES), which asks questions about caregiver self-efficacy related to understanding, navigating, and supporting their child's needs. The FES is an 24-question survey. Questions are measured on a five-point scale ranging from 1 (never) to 5 (very often). Possible survey scores can range from 24 to 120. Higher scores indicate greater self-perceived empowerment.
Child service access and utilization | Baseline to six-month follow-up
  Child service access and use will be measured using the Service Access and Utilization (SAU) questionnaire. The questionnaires asks about receipt of Part C early intervention services as well as private therapy services. Caregivers will complete the questionnaire at seven time points (approximately 15, 30, 45, 60, 90, 120, and 180 days following initial evaluation). At each time point, caregivers will endorse service milestones they have reached (e.g., scheduled an evaluation with the Part C service system, created an Individualized Family Service Plan, began services). We will calculate time to each milestone for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Warren, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- UC Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gangi DN, Corona L, Wagner L, Weitlauf A, Warren Z, Ozonoff S. In-home Tele-assessment for Autism in Toddlers: Validity, Reliability, and Caregiver Satisfaction with the TELE-ASD-PEDS. J Dev Behav Pediatr. 2025 Jun 17;46(3):e261-e268. doi: 10.1097/DBP.0000000000001358. PMID 40526421
- [Derived] Ozonoff S, Gangi D, Corona L, Foster T, Hill MM, Honaker M, Maqbool S, Ni R, Nicholson A, Parikh C, Stone C, Spitler AK, Swanson A, Vehorn A, Wagner L, Weitlauf A, Warren Z. Measuring Developmental Delays: Comparison of Parent Report and Direct Testing. J Autism Dev Disord. 2025 Dec;55(12):4492-4498. doi: 10.1007/s10803-024-06292-8. Epub 2024 Feb 26. PMID 38407697